CLINICAL TRIAL: NCT06554392
Title: Identification of Glutathione Peroxidase 4 in Detecting Ferroptosis in Ankylosing Spondylitis and Axial Psoriatic Arthritis Patients .
Brief Title: Identification of Serum Level of Glutathione Peroxidase 4
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Abdel Hakeem Abdullah Fahem, resident doctor, Assiut University
Other Study IDs: Glutathione Peroxidase 4
Record Dates: First submitted 2024-08-11; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Spondyloarthropathy
MeSH Terms: conditions — Spondylarthropathies | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ankylosing Spondylitis patients: Identification of Glutathione Peroxidase 4 in blood.
  Interventions: Diagnostic Test: Blood sample
- Axial Psoriatic Arthritis Patients: Identification of Glutathione Peroxidase 4 in blood.
  Interventions: Diagnostic Test: Blood sample
- healthy controls: Identification of Glutathione Peroxidase 4 in blood.
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample from each subject to detect Glutathione Peroxidase 4.

SUMMARY:
* Analysis of the level of glutathione peroxidase 4 (GPX4) in ankylosing spondylitis and axial psoriatic arthritis patients.
* The association of glutathione peroxidase 4 (GPX4) with disease activity and severity in ankylosing spondylitis and axial psoriatic arthritis patients.

DETAILED DESCRIPTION:
Ferroptosis, first reported by Dixon et al. in 2012, is a form of non-apoptotic cell death driven by iron-dependent lipid reactive oxygen species (ROS) and accelerated by the accumulation of lipid peroxides, ultimately leading to oxidative damage to phospholipid membranes and cell death .

Ferroptosis could be induced by iron metabolism disorder, lipid peroxidation accumulation, deficiency of glutathione (GSH) and inactivation of the antioxidant enzyme glutathione peroxidase 4 (GPX4).

The morphological features of ferroptotic cells manifest as an aberrant mitochondrial ultrastructure, including a reduction in mitochondrial volume, an increase in mitochondrial membrane density, and the disappearance of mitochondrial cristae in ferroptotic cells .

Recent studies have increasingly reported on complex associations between ferroptosis and the immune system . The regulatory activity of ferroptosis in immune function and inflammation is multifaceted and involves innate, acquired, and autoimmunity.

Accumulating evidence in recent times has shown an association of ferroptosis with the pathogenesis and development of autoimmune diseases .

Spondyloarthropathy comprises a group of chronic inflammatory rheumatic diseases, including ankylosing spondylitis, reactive arthritis (Reiter syndrome), arthritis or spondylitis associated with inflammatory bowel disease, and psoriatic arthritis, as well as undifferentiated spondyloarthritis. These afflictions predominantly affect the axial skeleton, causing pain and stiffness.

Currently, research on ferroptosis is still in its early stages; therefore, exploring the pathogenesis of ferroptosis and its role in various diseases, and proposing effective and targeted treatment methods have significant theoretical significance and practical value.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as ankylosing spondylitis according to ASAS criteria . [13]
* Patients diagnosed as psoriatic arthritis according to CASPAR criteria. [14]
* Age (>18).

Exclusion Criteria:

* Patient with other autoimmune Rheumatic diseases.
* patients with any of the following conditions: I) severe liver and kidney dysfunction; II) hematopoietic diseases; III) infectious diseases; IV) tumors; or V) other wasting diseases. [15]
* patients received certain drugs (for example, sulfasalazine, artemisinin, statins), and experimental reagents (such as erastin) .[16]

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from AS and axial psoriatic arthritis patients presented sequentially at the outpatient clinic and inpatient unit of the Department of Rheumatology, Rehabilitation and Physical Medicine. Faculty of Medicine .Assiut University.in addition to age and sex matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of the serum level of glutathione peroxidase 4 (GPX4) in ankylosing spondylitis and axial psoriatic arthritis patients. | baseline
  Analysis of the serum level of glutathione peroxidase 4 (GPX4) in ankylosing spondylitis and axial psoriatic arthritis patients to detect ferroptosis process in those patients.

SECONDARY OUTCOMES:
The association of glutathione peroxidase 4 (GPX4) with disease activity and severity in ankylosing spondylitis and axial psoriatic arthritis patients. | baseline
  The association of glutathione peroxidase 4 (GPX4) with disease activity and severity in ankylosing spondylitis and axial psoriatic arthritis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Abdelaziz, Prof., Study Director — Rheumatology,Rehabilition,Physical therapy Department ,Assiut university; Marwa Galal, Ass. Prof., Study Director — Rheumatology,Rehabilition,Physical therapy Department ,Assiut university; Nesreen Ibrahim, Dr, Study Director — Rheumatology,Rehabilition,Physical therapy Department ,Assiut university

REFERENCES:
- [Background] Dixon SJ, Lemberg KM, Lamprecht MR, Skouta R, Zaitsev EM, Gleason CE, Patel DN, Bauer AJ, Cantley AM, Yang WS, Morrison B 3rd, Stockwell BR. Ferroptosis: an iron-dependent form of nonapoptotic cell death. Cell. 2012 May 25;149(5):1060-72. doi: 10.1016/j.cell.2012.03.042. PMID 22632970
- [Background] Chen R, Zhu S, Zeng L, Wang Q, Sheng Y, Zhou B, Tang D, Kang R. AGER-Mediated Lipid Peroxidation Drives Caspase-11 Inflammasome Activation in Sepsis. Front Immunol. 2019 Aug 8;10:1904. doi: 10.3389/fimmu.2019.01904. eCollection 2019. PMID 31440260
- [Background] Yuan S, Wei C, Liu G, Zhang L, Li J, Li L, Cai S, Fang L. Sorafenib attenuates liver fibrosis by triggering hepatic stellate cell ferroptosis via HIF-1alpha/SLC7A11 pathway. Cell Prolif. 2022 Jan;55(1):e13158. doi: 10.1111/cpr.13158. Epub 2021 Nov 22. PMID 34811833
- [Background] Gao M, Yi J, Zhu J, Minikes AM, Monian P, Thompson CB, Jiang X. Role of Mitochondria in Ferroptosis. Mol Cell. 2019 Jan 17;73(2):354-363.e3. doi: 10.1016/j.molcel.2018.10.042. Epub 2018 Dec 20. PMID 30581146
- [Background] Chen X, Kang R, Kroemer G, Tang D. Ferroptosis in infection, inflammation, and immunity. J Exp Med. 2021 Jun 7;218(6):e20210518. doi: 10.1084/jem.20210518. Epub 2021 May 12. PMID 33978684